CLINICAL TRIAL: NCT04017494
Title: Validation of Cardiac Magnetic Resonance Sequences in Patients With Single Ventricles
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Barbara Burkhardt (Other)
Responsible Party: Sponsor-Investigator, Barbara Burkhardt, Principal Investigator, University Children's Hospital, Zurich
Organization: University Children's Hospital, Zurich (Other)
Other Study IDs: SV-CMR
Record Dates: First submitted 2019-07-08; First posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Single-ventricle
Keywords: Fontan; Congenital heart defects; Non-invasive cardiac imaging; Biomarkers
MeSH Terms: conditions — Univentricular Heart; Heart Defects, Congenital | interventions — Blood Specimen Collection; Hematocrit; Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single ventricle: Patients with single ventricle lesions
  Interventions: Diagnostic Test: Cardiac Magnetic Resonance Imaging; Diagnostic Test: Blood draw for hematocrit and heart failure biomarkers; Diagnostic Test: Cardiopulmonary exercise test; Diagnostic Test: Exhalomics; Diagnostic Test: Quality of life questionnaire

INTERVENTIONS:
Diagnostic Test: Cardiac Magnetic Resonance Imaging — Cardiac Magnetic Resonance Imaging (non-invasive, with i.v. application of contrast), awake or (if clinically indicated) in general anesthesia
Diagnostic Test: Blood draw for hematocrit and heart failure biomarkers — Approximately 10 ml of blood will be drawn before administration of contrast medium.
Diagnostic Test: Cardiopulmonary exercise test — In patients 8 years of age or older: on a cycle ergometer with breath-by-breath analysis, continuous ECG and SpO2 monitoring during exercise, after a baseline spirometry and bodyplethysmography
Diagnostic Test: Exhalomics — Measurement of exhaled molecules by mass spectrometry; patients breathe into a mouthpiece for 15 seconds 6 times (total time requirement: about 5 minutes)
Diagnostic Test: Quality of life questionnaire — Questionnaire to be filled out by the Patient regarding quality of life perception

SUMMARY:
Single ventricle defects make up the severe end of the congenital heart disease spectrum. The Fontan operation leads to a complete redirection of systemic venous blood outside of the heart and directly into the lungs. Patients with single ventricles suffer from multiple complications. Their survival has improved over the past decades, but is still severely compromised compared to the general population.

Their evaluation includes echocardiography and functional status by history and/or exercise testing. In longer intervals or if echocardiography does not allow visualization of all cardiovascular structures, cardiac magnetic resonance (CMR) is employed. Many patients also undergo more invasive cardiac catheterization.

In single ventricle patients, cardiac imaging has to address the questions of the patency of the Fontan pathways, i.e. all systemic veins, the Fontan conduit, and the pulmonary arteries, and of the function of the single ventricle (including myocardial function and valve function).

By using conventional imaging methods in Fontan patients, Ghelani et al. identified a CMR-based ventricular end-diastolic volume of > 125 ml/m2 and an echocardiographic global circumferential strain (GCS) value of higher than -17% to be strong predictors for a combined adverse outcome of death or heart transplantation. While interobserver reproducibility of single ventricle ejection fraction is similarly high by echocardiography, CMR is better in reliably measuring ventricular mass and diastolic volume and can provide additional information by MR feature tracking (strain), T1 mapping, and 4D flow measurements. Several substances that can be measured in the peripheral blood are being increasingly investigated as biomarkers of heart failure.

In conclusion, several advanced CMR sequences and new biomarkers have a potential role in the assessment and risk stratification of single ventricle patients. Every single published study has elucidated a particular use and aspect of these parameters, but broader correlations and prognostic values are still unclear.

The investigators hypothesize that myocardial strain (by feature tracking), myocardial fibrosis (by T1 mapping), and intracardiac flow disturbances (by 4D flow) along with biomarkers are diagnostic for single ventricle dysfunction and correlate with known prognostic factors.

This is a single center, prospective, observational cohort study. There will be no randomisation or blinding. Study setting: outpatients, cardiology clinic and radiology department, academic hospital. Every patient will be examined twice with a one-year interval (MR will only be repeated if clinically indicated).

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age with functionally single ventricle (patients under age 8 who need anesthesia for CMR will not be actively recruited. They may be approached to participate only if the anesthesia and CMR examination have been planned independently for clinical purposes)
* Written informed consent

Exclusion Criteria:

* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, inability to give assent or consent, etc. of the participant and/or his/her parents or legal caregivers
* MR-incompatible implanted or accidentally incorporated metal device or claustrophobia that prohibits use of magnetic resonance imaging (patient and guardians fill out a questionnaire).
* Pregnancy
* Participation in another study is not an exclusion criterion, e.g. in a therapeutic trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with single ventricle physiology
Sampling Method: Non-Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Strain correlation with ventricular volume | 1 year
  Strain correlation with ventricular volume measured by magnetic resonance imaging
Strain correlation with clinical parameters | 1 year
  Strain correlation with clinical parameters such as presence of arrhythmias on Holter-EKG, maximal oxygen consumption on cardio-pulmonary exercise testing (ml/(kg*min))

SECONDARY OUTCOMES:
T1 values compared to previously established normal cohort | 1 year
  T1 values compared to previously established normal cohort
Blood and exhaled biomarkers of heart failure correlation with T1 mapping | 1 year
  Blood and exhaled biomarkers of heart failure correlation with T1 mapping
Intraventricular blood flow correlation with cardiac function | 1 year
  Intraventricular blood flow correlation with cardiac ejection fraction measured by magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Barbara EU Burkhardt, MD, Principal Investigator — University of Zurich Children's Hospital
Locations (1):
- University Children's Hospital Zürich, Switzerland, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No